CLINICAL TRIAL: NCT02753842
Title: A Double-Blind, Single Center, Randomized 3-way Crossover Trial to Determine Pleasure for Fitted, Thin and Standard Condoms, and to Assess Clinical Failure for Vaginal and Anal Sex
Brief Title: Condom Performance in a Longitudinal Enhanced Assessment of User Experiences
Acronym: C-PLEASURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Global Protection Corp. (Industry)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Aaron Siegler, PhD, Emory University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB00083754
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: HIV
Keywords: Sexually Transmitted Infections; Condoms; Contraceptive Devices; HIV
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: We recruited 504 participants into the crossover trial. Participants were randomized into one of six sequences, each representing the order in which a participant would receive batches of five study condoms of a particular type.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In this closed label trial, study condoms were manufactured in plain foil packaging with identifying 2-digit random codes printed on each foil. Blinding of study staff was role-based; the study statistician and the principal investigator were blinded. To allow for blinded participants to identify preferred condoms, we provided condom sets in color-coded bags. We selected colors that could accommodate common forms of color vision deficiency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Fitted, Then Thin, Then Standard Condoms (Experimental): Participants first received 5 fitted condoms, and had a period of 2-4 weeks to use them. They then received 5 thin condoms, and had a period of 2-4 weeks to use them. They then received 5 standard condoms, and had a period of 2-4 weeks to use them.
  Interventions: Device: 5 Fitted Condoms, 5 Thin Condoms, 5 Standard Condoms
- Fitted, Then Standard, Then Thin Condoms (Experimental): Participants first received 5 fitted condoms, and had a period of 2-4 weeks to use them. They then received 5 standard condoms, and had a period of 2-4 weeks to use them. They then received 5 thin condoms, and had a period of 2-4 weeks to use them.
  Interventions: Device: 5 Fitted Condoms, 5 Thin Condoms, 5 Standard Condoms
- Thin, Then Fitted, Then Standard Condoms (Experimental): Participants first received 5 thin condoms, and had a period of 2-4 weeks to use them. They then received 5 fitted condoms, and had a period of 2-4 weeks to use them. They then received 5 standard condoms, and had a period of 2-4 weeks to use them.
  Interventions: Device: 5 Fitted Condoms, 5 Thin Condoms, 5 Standard Condoms
- Thin, Then Standard, Then Fitted Condoms (Experimental): Participants first received 5 thin condoms, and had a period of 2-4 weeks to use them. They then received 5 standard condoms, and had a period of 2-4 weeks to use them. They then received 5 fitted condoms, and had a period of 2-4 weeks to use them.
  Interventions: Device: 5 Fitted Condoms, 5 Thin Condoms, 5 Standard Condoms
- Standard, Then Fitted, Then Thin Condoms (Experimental): Participants first received 5 standard condoms, and had a period of 2-4 weeks to use them. They then received 5 fitted condoms, and had a period of 2-4 weeks to use them. They then received 5 thin condoms, and had a period of 2-4 weeks to use them.
  Interventions: Device: 5 Fitted Condoms, 5 Thin Condoms, 5 Standard Condoms
- Standard, Then Thin, Then Fitted Condoms (Experimental): Participants first received 5 standard condoms, and had a period of 2-4 weeks to use them. They then received 5 thin condoms, and had a period of 2-4 weeks to use them. They then received 5 fitted condoms, and had a period of 2-4 weeks to use them.
  Interventions: Device: 5 Fitted Condoms, 5 Thin Condoms, 5 Standard Condoms

INTERVENTIONS:
Device: 5 Fitted Condoms, 5 Thin Condoms, 5 Standard Condoms — Fitted condoms are available in 56 sizes based on combinations of length (approximately 10mm increments) and circumference (approximately 2 mm increments). Fitted condom thickness is 70 microns ± 10 microns. Appropriate condom size is user-determined with a paper template fitting tool graduated with non-sequential numbering and lettering for maximum privacy. Participants also received ten plain foil packets of 10ml commercially available condom-compatible water-based lubricant.
  Thin condoms have dimensions of 185mm ± 10mm length, 53mm ± 2mm width, and 50 microns ± 5 microns thick. Participants also received ten plain foil packets of 10ml commercially available condom-compatible water-based lubricant.
  Standard condoms have dimensions of 185mm ± 10mm length, 53mm ± 2mm width, and 70 microns ± 10 microns thick. Participants also received ten plain foil packets of 10ml commercially available condom-compatible water-based lubricant.

SUMMARY:
This study will enroll 252 men who have sex with men (MSM) and 252 men who have sex with women (MSW) in a double-blind, three-way randomized crossover trial with conditions of fitted, thin, and standard condoms. The study will provide fitted condoms in 56 sizes based on combinations of length (approximately 10 mm increments) and circumference (approximately 2 mm increments), with user-determined size based on a paper template measurement instrument.

Participants will be randomly assigned to the sequence in which the crossover intervention conditions (fitted, thin, and standard condoms) occur, with five study condoms provided for each condition. Participants will attend at least four, and up to seven, biweekly study visits.

DETAILED DESCRIPTION:
Study objectives are to establish label indications for pleasure and patient preference for fitted condoms, establish label indication for anal sex for fitted, thin, and standard condoms, and establish a label indication for decreased clinical failure of fitted condoms for anal sex.

The study will enroll 252 MSM and 252 men who sex with women (MSW) into a double-blind, three-way randomized crossover trial with conditions of fitted, thin, and standard condoms. For MSM enrolled in the trial we will assess outcomes based on anal sex, and for MSW we will assess outcomes based on vaginal sex. The study will provide fitted condoms in 56 sizes based on combinations of length (approximately 10 mm increments) and circumference (approximately 2 mm increments), with user-determined size based on a paper template measurement instrument.

For purposes of this study, a "standard" condom is defined by dimensions commonly sourced by the United Nations Population Fund (UNFPA) and United States Agency for International Development (USAID), which procures the majority of the world's condoms. These dimensions are 185mm ± 10mm length, 53mm ± 2mm width, and 70 microns ± 10 microns thick. "Thin" condoms for this study will be of identical width and length to "standard", but 50 microns ± 5 microns thick. Fitted condoms will be produced in a range of sizes with thickness of 70 microns ± 10 microns, with a participant's fitted size as determined by their use of a fitting system consisting of a paper template graduated with non-sequential numbering and lettering. Condoms will be manufactured using the same latex formulation and silicone lubricants (approximately 400mg per condom), and with similar parallel wall designs.

Every participant in the trial will receive a set of five fitted condoms (fitted condition), a set of five thin condoms (thin condition), and a set of five standard condoms (standard condition) over a series of study visits. Event-level data based on a home coital log will be collected regarding pleasure and total clinical failure, and data regarding overall condom preference will be collected at the final study visit. Participants will be randomly assigned to the sequence in which the crossover intervention conditions (fitted, thin, and standard) occur. Each participant will attend at least four, and up to seven, biweekly study visits. Participants will be given up to four weeks to use each study condom set; after 4 weeks with a set of condoms, participants will be automatically crossed over into the next study condition. If all condoms are used within the first two weeks, participants will crossover to the next randomized condition.

Participants will be blinded, with all condoms produced in plain foils with two-digit identifying codes, and role-based blinding will be conducted for study staff with the statistician and PI blinded. Participants will be trained in appropriate condom use, fitted condom sizing, study instructions such as only using study lubricant, and daily coital log completion. Participants will complete mobile-optimized, web-based home coital logs as soon as possible following any vaginal or anal sex acts. To assist participants in timely completion, there will be a daily check-in through Short Message Service (SMS) (via text message) with a reminder initiated if no sexual event has been recently reported. The coital log will include outcome measures for pleasure and for condom failure. The final visit survey will measure overall condom preference.

ELIGIBILITY:
Inclusion Criteria:

* Lives in or near Atlanta metropolitan statistical area (MSA)
* Plans to be in Atlanta for the majority of the 12 weeks of enrollment
* Able to independently complete survey instruments in English
* Male sex at birth
* Currently identifies as male
* For MSM, self-report to have only had sex with men in the past four weeks
* For MSM, self-report intends to have sex only with men in the next 12 weeks
* For MSW, self-report to have only had sex with women in the past four weeks
* For MSW, self-report intends to have sex only with women in the next 12 weeks
* Self-report at least 1 anal (MSM) or vaginal (MSW) sex act in the past four weeks
* For MSM, self-reports an insertive role in the past four weeks
* Willing and able to have sex using a latex condom provided by study
* Consistently able to maintain an erection while using condoms
* Willing to provide at least two means of contact
* Willing to only use lubricant provided by study
* Willing to use a fitting tool to determine penile dimensions

Exclusion Criteria:

* Self-report transgender sex partners in the past four weeks
* Plans to not have sex in the next four weeks
* For MSW, report that current partner is currently pregnant
* For MSW, report that current partner desires to become pregnant currently or in the next 12 weeks
* Allergic to latex
* Current partner(s) allergic to latex
* Genital piercings
* For MSW, female current partner(s) has (have) vaginal piercings
* For MSM, male current partner(s) has (have) anal piercings
* Current partner(s) known to be HIV-positive
* Self-report presence of sexually transmitted infections, including HIV
* Confirmed HIV positive at baseline
* Allergic to water-based lubricant
* Current partner(s) allergic to water-based lubricant

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 504 (Actual)
Dates: Start 2016-05; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron J Siegler, PhD, Study Director — Emory University

REFERENCES:
- [Background] Siegler AJ, Rosenthal EM, Sullivan PS, Ahlschlager L, Kelley CF, Mehta CC, Moore RH, Rosenberg ES, Cecil MP. Double-Blind, Single-Center, Randomized Three-Way Crossover Trial of Fitted, Thin, and Standard Condoms for Vaginal and Anal Sex: C-PLEASURE Study Protocol and Baseline Data. JMIR Res Protoc. 2019 Apr 23;8(4):e12205. doi: 10.2196/12205. PMID 31012862
- [Result] Siegler AJ, Rosenthal EM, Sullivan PS, Christina Mehta C, Moore RH, Ahlschlager L, Kelley CF, Rosenberg ES, Cecil MP. Levels of clinical condom failure for anal sex: A randomized cross-over trial. EClinicalMedicine. 2019 Oct 31;17:100199. doi: 10.1016/j.eclinm.2019.10.012. eCollection 2019 Dec. PMID 31891134

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in Atlanta, GA from May 19, 2016 - May 2, 2017. Recruitment was predominantly through electronic advertising and paper signs posted at venues such as college campuses.
Pre-assignment Details: We recruited 504 participants into the crossover trial. Participants were randomized into one of six sequences, each representing the order in which a participant would receive batches of five study condoms of a particular type.
Period: First Follow-Up (Set of Condoms)
Arm/Group | Fitted, Then Thin, Then Standard Condoms | Fitted, Then Standard, Then Thin Condoms | Thin, Then Fitted, Then Standard Condoms | Thin, Then Standard, Then Fitted Condoms | Standard, Then Fitted, Then Thin Condoms | Standard, Then Thin, Then Fitted Condoms
Started | 85 | 84 | 85 | 83 | 83 | 84
Completed | 75 | 76 | 76 | 81 | 76 | 79
Not Completed | 10 | 8 | 9 | 2 | 7 | 5
Period: Second Follow-Up (Set of Condoms)
Arm/Group | Fitted, Then Thin, Then Standard Condoms | Fitted, Then Standard, Then Thin Condoms | Thin, Then Fitted, Then Standard Condoms | Thin, Then Standard, Then Fitted Condoms | Standard, Then Fitted, Then Thin Condoms | Standard, Then Thin, Then Fitted Condoms
Started | 75 | 76 | 76 | 81 | 76 | 79
Completed | 71 | 71 | 71 | 76 | 75 | 72
Not Completed | 4 | 5 | 5 | 5 | 1 | 7
Period: Third Follow-Up (Set of Condoms)
Arm/Group | Fitted, Then Thin, Then Standard Condoms | Fitted, Then Standard, Then Thin Condoms | Thin, Then Fitted, Then Standard Condoms | Thin, Then Standard, Then Fitted Condoms | Standard, Then Fitted, Then Thin Condoms | Standard, Then Thin, Then Fitted Condoms
Started | 71 | 71 | 71 | 76 | 75 | 72
Completed | 65 | 66 | 68 | 70 | 71 | 69
Not Completed | 6 | 5 | 3 | 6 | 4 | 3

BASELINE CHARACTERISTICS:
Population: All participants completed baseline data collection.
Groups:
- Fitted, Then Thin, Then Standard Condoms: Fitted, Then Thin, Then Standard Condoms.
- Fitted, Then Standard, Then Thin Condoms: Fitted, Then Standard, Then Thin Condoms.
- Thin, Then Fitted, Then Standard Condoms: Thin, Then Fitted, Then Standard Condoms.
- Thin, Then Standard, Then Fitted Condoms: Thin, Then Standard, Then Fitted Condoms.
- Standard, Then Fitted, Then Thin Condoms: Standard, Then Fitted, Then Thin Condoms.
- Standard, Then Thin, Then Fitted Condoms: Standard, Then Thin, Then Fitted Condoms.
- Total: Total of all reporting groups
Arm/Group | Fitted, Then Thin, Then Standard Condoms | Fitted, Then Standard, Then Thin Condoms | Thin, Then Fitted, Then Standard Condoms | Thin, Then Standard, Then Fitted Condoms | Standard, Then Fitted, Then Thin Condoms | Standard, Then Thin, Then Fitted Condoms | Total
Number analyzed (Participants) | 85 | 84 | 85 | 83 | 83 | 84 | 504
Age, Customized [Count of Participants; unit: Participants]
  < 20 years | 9 | 11 | 9 | 8 | 15 | 4 | 56
  20-24 years | 28 | 25 | 29 | 29 | 21 | 26 | 158
  25-29 years | 16 | 19 | 22 | 20 | 24 | 22 | 123
  30-39 years | 23 | 20 | 16 | 19 | 15 | 15 | 108
  40-54 years | 9 | 9 | 9 | 7 | 8 | 17 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 85 | 84 | 85 | 83 | 83 | 84 | 504
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 7 | 13 | 12 | 11 | 6 | 13 | 62
  White non-Hispanic | 45 | 40 | 44 | 32 | 40 | 40 | 241
  African-American non-Hispanic | 18 | 23 | 19 | 25 | 23 | 23 | 131
  Other non-Hispanic | 15 | 8 | 10 | 14 | 14 | 8 | 69
  Prefer not to answer, non-Hispanic | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 85 | 84 | 85 | 83 | 83 | 84 | 504

OUTCOME MEASURES:

1. Primary Outcome: Sexual Pleasure Scale Score for Fitted Versus Standard Condoms
Description: Our aim was to compare fitted condoms with standard condoms regarding levels of reported pleasure, as determined by rating per condom use event. The sexual pleasure scale for this study was developed and validated by the study team (Siegler et. al., Arch Sex Behav. 2018 Aug; 47(6): 1745-1754), and is titled event-level, male sexual pleasure scale (EMSEXpleasure). The scale comprises 11 items with sliding scale response scores. Pleasure scale measurement was assessed with a mobile-optimized, web-based home daily coital log, completed following each coital event. The minimum scale score was zero, the maximum was 100. Higher values indicate greater pleasure.
  We assessed the difference in mean scores of pleasure for fitted condoms versus standard condoms.
Time Frame: Up to 12 weeks
Population: The analysis is comprised of pleasure scale scores completed after each sex act, when a study condom was used.
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Sex acts with study condoms
Groups:
- Fitted Condoms: Participants received all conditions (fitted condoms, thin condoms, and standard condoms), with the order in which condoms are received based on permuted block randomization.
- Standard Condoms: Participants will receive all conditions (fitted condoms, thin condoms, and standard condoms), with the order in which condoms are received based on permuted block randomization.
Arm/Group | Fitted Condoms | Standard Condoms
Number analyzed (Participants) | 485 | 485
Number analyzed (Sex acts with study condoms) | 4740 | 4740
score on a scale | 71.52 (0.77) | 70.13 (0.78)
Statistical Analysis 1: Comparison: Fitted Condoms vs Standard Condoms; Comparing fitted to standard condoms, the null hypothesis was no difference in pleasure; Test type: Superiority; p < 0.05, Mixed Models Analysis — The a priori threshold was p<0.05; Mean Difference (Final Values) = 1.39, 95% CI 2-sided [0.52 to 2.26]

2. Primary Outcome: Percent of Participants Preferring Fitted Condoms to Standard Condoms
Description: Our aim was to compare fitted condoms with standard condoms regarding preference, as determined by ranking of the two conditions at the study conclusion.
  Condom preference was determined by participants selecting a preference for fitted or standard condoms at the study conclusion. The measure used assessed a blinded preference, referring to the color assigned to the condom type rather than the type of condom by name.
Time Frame: Up to 12 weeks
Population: Participants who used at least one fitted and one standard condom
Measure: Number (95% Confidence Interval); unit: % of participants prefer fitted condoms
Groups:
- Condom Preference (Binary): Preference for fitted or standard condoms at the end of the study. Participants were blinded to condom type.
Arm/Group | Condom Preference (Binary)
Number analyzed (Participants) | 371
% of participants prefer fitted condoms | 53.0 [47.9 to 58.1]
Statistical Analysis 1: Comparison: Condom Preference (Binary); A single item assessed whether participants preferred fitted condoms or standard condoms at the end of the study (the item word viewed by participants used the blinded identifiers of each condom type); Test type: Superiority; p > 0.05, Mixed Models Analysis; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.92 to 1.38]

3. Primary Outcome: Clinical Condom Failure for Anal Sex
Description: Our aim was to assess for fitted, thin, and standard condoms the total clinical failure rate of each type of condom for anal sex among MSM relative to the 5% failure cut-point previously used by the United States Food and Drug Administration (FDA). Clinical condom failure (condom breakage and slippage) was assessed by questions from the International Organization for Standardization (ISO), with a mobile-optimized, web-based home daily coital log completed following each coital event. Clinical failure was calculated according to ISO guidance.
Time Frame: Up to 12 weeks
Population: Participants who used at least one condom during the study
Measure: Count of Units; unit: Condoms
Units Other Than Participants: Condoms
Groups:
- Fitted Condoms: Fitted condoms used for anal sex
- Thin Condoms: Thin condoms used for anal sex
- Standard Condoms: Standard condoms used for anal sex
Arm/Group | Fitted Condoms | Thin Condoms | Standard Condoms
Number analyzed (Participants) | 216 | 210 | 206
Number analyzed (Condoms) | 813 | 788 | 750
Condoms | 5 | 6 | 5

4. Primary Outcome: Clinical Condom Failure of Fitted Condoms Compared to Standard Condoms for Anal Sex
Description: Our aim was to compare fitted condoms with standard condoms regarding total clinical failure for anal sex among MSM. Clinical condom failure (condom breakage and slippage) was assessed based on questions suggested by the International Organization for Standardization (ISO) and with a mobile-optimized, web-based home daily coital log completed following each coital event. Clinical failure was calculated according to ISO guidance.
Time Frame: Up to 12 weeks
Population: Persons contributing data regarding performance of at least one condom in the condition.
Measure: Count of Units; unit: Condoms
Units Other Than Participants: Condoms
Groups:
- Fitted Condoms Used for Anal Sex: Fitted condom clinical failure when used for anal sex
- Standard Condoms Used for Anal Sex: Standard condom clinical failure when used for anal sex
Arm/Group | Fitted Condoms Used for Anal Sex | Standard Condoms Used for Anal Sex
Number analyzed (Participants) | 216 | 206
Number analyzed (Condoms) | 813 | 750
Condoms | 5 | 5
Statistical Analysis 1: Comparison: Fitted Condoms Used for Anal Sex vs Standard Condoms Used for Anal Sex; We assessed clinical condom failure for anal sex, comparing anal sex acts with fitted condoms to anal sex acts with standard condoms; Test type: Superiority; p > 0.05, logistic mixed effects model; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.27 to 3.24]

5. Secondary Outcome: Sexual Pleasure Scale Score for Thin Versus Standard Condoms
Description: This secondary outcome sought to compare thin condoms with standard condoms regarding levels of reported pleasure, as determined by rating per condom use event. The sexual pleasure scale for this study was developed and validated by the study team (Siegler et. al., Arch Sex Behav. 2018 Aug; 47(6): 1745-1754), and is titled event-level, male sexual pleasure scale (EMSEXpleasure). The scale comprises 11 items with sliding scale response scores. Pleasure scale measurement was assessed with a mobile-optimized, web-based home daily coital log, completed following each coital event. The minimum scale score was zero, the maximum was 100. Higher values indicate greater pleasure.
  We assessed the difference in mean scores of pleasure for thin condoms versus standard condoms.
Time Frame: Up to 12 weeks
Population: The analysis is comprised of pleasure scale scores completed after each sex act, when a study condom was used.
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Sex acts with study condoms
Groups:
- Thin Condoms: Participants received all conditions (fitted condoms, thin condoms, and standard condoms), with the order in which condoms are received based on permuted block randomization.
Arm/Group | Thin Condoms | Standard Condoms
Number analyzed (Participants) | 485 | 485
Number analyzed (Sex acts with study condoms) | 4740 | 4740
score on a scale | 71.19 (0.77) | 70.13 (0.78)
Statistical Analysis 1: Comparison: Thin Condoms vs Standard Condoms; Comparing thin to standard condoms, the null hypothesis was no difference in pleasure; Test type: Superiority; p < 0.05, Mixed Models Analysis — The a priori threshold was p<0.05; Median Difference (Final Values) = 1.06, 95% CI 2-sided [0.18 to 1.94]

ADVERSE EVENTS:
Time Frame: The period of study participation, ranging from 0-12 weeks.
Description: We used standard definitions for adverse events
Groups:
- Fitted Condoms: Fitted condoms are available in 56 sizes based on combinations of length (approximately 10mm increments) and circumference (approximately 2 mm increments). Fitted condom thickness is 70 microns ± 10 microns. Appropriate condom size is user-determined with a paper template fitting tool graduated with non- sequential numbering and lettering for maximum privacy. Participants also received ten plain foil packets of 10ml commercially available condom-compatible water-based lubricant.
- Thin Condoms: Thin condoms have dimensions of 185mm ± 10mm length, 53mm ± 2mm width, and 50 microns ± 5 microns thick. Participants also received ten plain foil packets of 10ml commercially available condom-compatible water-based lubricant.
- Standard Condoms: Standard condoms have dimensions of 185mm ± 10mm length, 53mm ± 2mm width, and 70 microns ± 10 microns thick. Participants also received ten plain foil packets of 10ml commercially available condom-compatible water-based lubricant.
Arm/Group | Fitted Condoms | Thin Condoms | Standard Condoms
All-Cause Mortality (participants affected / at risk) | 0/468 | 0/469 | 0/464
Serious Adverse Events (participants affected / at risk) | 0/468 | 0/469 | 0/464
Other Adverse Events (participants affected / at risk) | 9/468 | 11/469 | 6/464
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fitted Condoms (N=468) | Thin Condoms (N=469) | Standard Condoms (N=464)
Symptomatic STI or recent STI diagnosis (Investigations) | 3 (3) | 4 (4) | 2 (2)
Condom- or lube-related discomfort (Investigations) | 4 (4) | 7 (7) | 4 (4)
Partner discomfort with lubricant (Investigations) | 1 (1) | 0 (0) | 0 (0)
Partner Urinary Tract Infection (Investigations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-12-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT02753842/Prot_000.pdf
  • Informed Consent Form (2016-06-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT02753842/ICF_001.pdf
  • Statistical Analysis Plan (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT02753842/SAP_002.pdf